CLINICAL TRIAL: NCT03712891
Title: Evaluation of Providing Coffee to Patients Postoperatively to Decrease Length of Stay in the PACU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Principal Investigator, Rachel Baker, Nurse Researcher, TriHealth Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-050
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-10

CONDITIONS: PACU Length of Stay; Postoperative Nausea; Postoperative Vomiting; Patient Satisfaction
Keywords: PACU length of stay; coffee
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Patient Satisfaction | interventions — Coffee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients receiving coffee postoperatively (Experimental): Patients who self-identify as coffee drinkers and receive coffee postoperatively
  Interventions: Dietary Supplement: Coffee
- Patients not receiving coffee postoperatively (No Intervention): Patients who self-identify as coffee drinkers and do not receive coffee postoperatively

INTERVENTIONS:
Dietary Supplement: Coffee — Patients will receive coffee in a Styrofoam cup at a temperature of 125 degree Fahrenheit or less. Coffee will be offered to the patient in the PACU once the patient's gag reflex has been restored following their procedure. Volume of estimated coffee consumption will be measured using a sample scale (with a maximum of 300mL of coffee offered)
  Arms: Patients receiving coffee postoperatively

SUMMARY:
The purpose of the study is to determine if providing coffee to patients who self-identify as coffee drinkers postoperatively will decrease the length of stay in the post-anesthesia care unit (PACU).

DETAILED DESCRIPTION:
Decreasing the length of stay in PACU for surgical patient is a pertinent outcome. The shorter length of stay can achieve higher patient engagement scores, while simultaneously increasing the productivity of the unit. This is achieved by making more beds available for new patients coming from the operating room (OR). One thought was that coffee would benefit the investigator's patients experience through a number of pathways. Initially, the stimulant effect of coffee would create a more alert patient. A more alert patient is more likely to comprehend home care instruction and be ready for discharge earlier. Coffee is often used as a remedy for morning sickness. Ideally the act of drinking coffee or even smelling the coffee may decrease the occurrence of Post-Operative Nausea and Vomiting (PONV) in investigator's patient population. Finally, patients frequently state that the inability to drink their morning coffee is often more difficult than not being able to eat prior to surgery. By allowing those to drink coffee in PACU this would make the patient feel that they are being cared for on an emotional level, in addition to a physical level.

ELIGIBILITY:
Inclusion criteria:

1. 18 years old or older
2. Admitted to Bethesda North Minimally Invasive Surgery Center
3. Reports to consume at least one cup of coffee a day for at least 5 days in a week

Exclusion Criteria

1. History of PONV
2. Pre-existing cardiac arrhythmias
3. History of seizure disorder
4. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Ballhaus, BSN, RN, Principal Investigator — TriHealth Inc.
Locations (1):
- Bethesda North Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Receiving Coffee Postoperatively | Patients Not Receiving Coffee Postoperatively
Started | 89 | 89
Completed | 89 | 89
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Receiving Coffee Postoperatively | Patients Not Receiving Coffee Postoperatively | Total
Number analyzed (Participants) | 89 | 89 | 178
Age, Customized [Count of Participants; unit: Participants]
  18 years or older | 89 | 89 | 178
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Did not collect
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 89 | 89 | 178

OUTCOME MEASURES:

1. Primary Outcome: PACU Length of Stay
Description: Post-anesthesia Care Unit length of stay
Time Frame: 6 hours
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Patients Receiving Coffee Postoperatively | Patients Not Receiving Coffee Postoperatively
Number analyzed (Participants) | 89 | 89
minutes | 82 (5.13) | 76 (5.13)
Statistical Analysis 1: Comparison: Patients Receiving Coffee Postoperatively; Test type: Other — t-test; p = 0.12, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Patient level: Less than 6 hours Study level: During length of study
Arm/Group | Patients Receiving Coffee Postoperatively | Patients Not Receiving Coffee Postoperatively
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/89
Other Adverse Events (participants affected / at risk) | 0/89 | 0/89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT03712891/Prot_SAP_000.pdf